CLINICAL TRIAL: NCT05147441
Title: Evaluating the Efficacy of Obturator Cryoneurotomy for Hip Adductor Spasticity
Brief Title: Obturator Cryoneurotomy for Hip Adductor Spasticity
Status: Recruiting | Type: Observational
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Mahdis Hashemi, Research Assistant, Vancouver Island Health Authority
Other Study IDs: H21-01646
Record Dates: First submitted 2021-11-02; First posted 2021-12-07 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Spasticity, Muscle
Keywords: spasticity; Cryoneurotomy; Hip adductors; Range of motion
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to measure the effects of obturator nerve cryoneurotomy, on clinical measures in adult (ages 19+) and paediatric (ages 12-18) patients with hip adductor spasticity, who will receive this procedure as a part of their treatment based on the spasticity treatment available guidelines. The results will provide us valuable information like how long cryoneurotomy is effective, before regeneration happens

DETAILED DESCRIPTION:
Hip adductor spasticity is a common affliction amongst patients with disorders of the central nervous system. Spasticity affects as much as 60% of people with cerebral palsy, and up to 97% of patients with MS. Spasticity can be detrimental to gait, leading to lowered walking velocity, lack of stability and more frequent falls in conditions of the central nervous system, like cerebral palsy . Hip adductor spasticity can make it difficult for one to part their knees sufficiently to perform personal hygiene and can lead to extreme difficulties dressing and performing other activities of daily living. A lack of ability to perform activities of daily living leads to lessened independence. In this study, we will measure the efficacy of obturator cryoneurotomy for patients with spastic hip adduction as an alternative approach to more invasive, complicated and costly treatments.

Research Design

This project constitutes a single-centre, prospective cohort study. Data collection will occur at the Victoria General Hospital (VGH) multidisciplinary spasticity clinic, consisting of physiatrists, an orthopedic surgeon and physiotherapists. Patients with spasticity are referred to this clinic for different procedures including cryoneurotomy. This multidisciplinary spasticity clinic offers various treatments to spastic patients, including botulinum toxin injection, bracing, consultations for surgery or neurotomy. All procedures are offered to each patient. Most of the patients in the study will have already had Botox and bracing, or even neurotomy. As of yet all patients have had botulinum injections and bracing before cryoneurotomy. This study will not interfere or change the patients' medical care, and we will do the assessments for the patients who are already candidates for this procedure as a part of their treatment, besides other provided medical cares and have been accepted to receive that.

Patients who are already candidates for cryoneurotomy as a part of their treatment, will be invited to have an extra ten-meter walk test. All measures are part of the standard clinical assessment, except the 10 meter-walk test. The spasticity degree and range of motion will be measured for both limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Will have cryoneurotomy as part of their standard treatment for spastic hip adductors in VGH spasticity multidisciplinary clinic.
2. Are at least 12 years of age at the time of the procedure.
3. Have the ability to attend testing sessions, comply with testing protocols and provide written informed consent.
4. Are able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).

Exclusion Criteria:

1. Have a history of previous nerve procedures such as chemical neurolysis with alcohol, cryoneurotomy, or any surgery to the obturator nerve.
2. Have any other neurological pathology different from that responsible for the spasticity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are at least 12 years old and will have Cryoneurotomy as a part of their provided medical care will be asked to be enrolled in the study. All patients will be recruited through multidisciplinary spasticity clinic in Victoria General Hospital where spastic patients are referred to this center routinely.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The degree of changes in hip abductors' active range of motion. | measurement will be done at baseline, 1 month after having Cryoneurotomy and then every 3 months up to one year.
  any changes in active passive hip abduction range of motion will be measured by trained examiners with a standard goniometer.
The degree of changes in hip abductors' maximum passive range of motion. | measurement will be done at baseline, 1 month after having Cryoneurotomy and then every 3 months up to one year.
  any changes in maximum passive hip abduction range of motion will be measured by trained examiners with a standard goniometer
The degree of changes in hip abductors' spasticity | measurement will be done at baseline, 1 month after having Cryoneurotomy and then every 3 months up to one year.
  any changes in hip abduction will be measured based on Modified Ashworth Scale, which has 6 scores (from 0 which means no spasticity to 4 which means the highest degree of the spasticity).
The degree of changes in inter knees distance at maximum passive hip abduction range of motion | It will be done at baseline, 1 month after cryoneurotomy and then every 3 months up to 12 months
  The measurement will be done by measure tape and based on centimetre scale

SECONDARY OUTCOMES:
Any changes in the ability to perform hygienic care related to degree of adductor muscles spasticity | The assessment will be done at baseline, 1 month after cryoneurotomy and then every 3 months up to one year.
  The assessment will be based on a four-point scale: 0 means relatively easy and 3 means with severe difficulty (Viel et al.,2002)
Any changes in 10-meter walk test. | The assessment will be done at baseline, 1 month after cryoneurotomy and then every 3 months up to one year.
  Patients will be asked to walk in a designed area for 10 meter and twice. the result will be average time of 2 rounds and will be recorded as second.
Any changes in patients' gait based on the physician's observation and the patient's perception. | The assessment will be done at baseline, 1 month after cryoneurotomy and then every 3 months up to one year.
  The gait will be scored based on a 4-point scale: 0 will be assigned to patients with no difficulty in walking and 3 will be assigned to the patients who are unable to walk (Viel et al.,2002)
Any changes in degree of pain if they have any. | The assessment will be done at baseline, 1 month after cryoneurotomy and then every 3 months up to one year.
  Patients will be asked if they have any related pain and to score it based on 10-point scale, which 0means no pain and 10 means the worst pain that they ever experienced
Patients satisfaction in achieving their goals after the procedure as assessed by Goal Attainment Scale (Turner-Stokes, 2009). | The follow up will be done up to one year.
  Based on this scale participants will be asked for 3 main goals that they desire to achieve after the intervention. The baseline score will be (-1) and they will be interviewed again at 6 and 12 months, to record how they reported their achievement. The scores of (-2), (-0.5), (0), (+1) and (+2) will be assigned if they feel that their condition is worst than before, better but not as good as expected, as expected, better than expected and much better than expected. All goals will be weighted equally, and final score will be calculated based on the available formula, in each session. The higher score is presenting of better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes MP, Kent RM, Semlyen JK, McMullen KM. Spasticity in multiple sclerosis. Neurorehabil Neural Repair. 2003 Mar;17(1):66-70. doi: 10.1177/0888439002250449. PMID 12645447
- [Background] Tugui RD, Antonescu D. Cerebral palsy gait, clinical importance. Maedica (Bucur). 2013 Sep;8(4):388-93. PMID 24790675
- [Background] Mlinac ME, Feng MC. Assessment of Activities of Daily Living, Self-Care, and Independence. Arch Clin Neuropsychol. 2016 Sep;31(6):506-16. doi: 10.1093/arclin/acw049. Epub 2016 Jul 29. PMID 27475282
- [Background] Viel EJ, Perennou D, Ripart J, Pelissier J, Eledjam JJ. Neurolytic blockade of the obturator nerve for intractable spasticity of adductor thigh muscles. Eur J Pain. 2002;6(2):97-104. doi: 10.1053/eujp.2001.0269. PMID 11900470
- [Background] Turner-Stokes L. Goal attainment scaling (GAS) in rehabilitation: a practical guide. Clin Rehabil. 2009 Apr;23(4):362-70. doi: 10.1177/0269215508101742. Epub 2009 Jan 29. PMID 19179355

DOCUMENTS (3):
  • Informed Consent Form: Adult consent form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05147441/ICF_000.pdf
  • Informed Consent Form: Teen Assent form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05147441/ICF_001.pdf
  • Informed Consent Form: Kids Assent form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05147441/ICF_002.pdf